CLINICAL TRIAL: NCT03271515
Title: Phase I Study of T Cells Expressing an Anti-CD19 and Anti-CD20 Bispecific Chimeric Receptor in Patients With B Cell Malignancies
Brief Title: Immunotherapy With Bispecific CAR-T Cells for B-Cell Lymphoma, ALL and CLL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Doing Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Doing-006
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Leukemia; Lymphoma
Keywords: leukemia; lymphoma; CAR-T; bispecific; CD20; CD19
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (No Intervention): patients accept conventional radioactive and chemical therapy.
- anti-CD19 anti-CD20 Bispecific CAR-T (Experimental): patients accept transfusion of anti-CD19 anti-CD20 Bispecific CAR-T cells.
  Interventions: Biological: anti-CD19 anti-CD20 Bispecific CAR-T

INTERVENTIONS:
Biological: anti-CD19 anti-CD20 Bispecific CAR-T — patients accept transfusion of anti-CD19 anti-CD20 Bispecific CAR-T cells.
  Arms: anti-CD19 anti-CD20 Bispecific CAR-T

SUMMARY:
This study aims to evaluate the safety, efficacy and duration of response of anti-CD19 anti-CD20 Bispecific Chimeric Antigen Receptor (CAR) redirected autologous T-cells in patients with high risk, relapsed CD19+ and CD20+ haematological malignancies.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product named CD19 CD20 Chimeric Antigen Receptor (CAR) T-cells (CD19 CAR T-cells) in patients with high risk, relapsed CD19+ and CD20+haematological malignancies (Leukemia and lymphoma). Following informed consent and registration to the trial, patients will undergo an unstimulated leukapheresis for the generation of the CD19 CD20 CAR T-cells. Patients will receive the CD19 CD20 CAR T-cells following lymphodepleting chemotherapy. The study will evaluate the safety, efficacy and duration of response of the CD19 CD20 CAR T-cells in patients with high risk relapsed CD19+ malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B cell derived acute lymphoblastic leukemia(ALL), chronic lymphoblastic leukemia(CLL) and non-hodgkin lymphoma.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 18 years to 70 years.
5. CD19 or CD20 expression must be detected on greater than 15% of the malignant cells by immunohistochemistry or greater than 30% by flow cytometry.
6. Patients who have failed at least one line of a standard treatment.
7. No serious mental disorder.
8. Patients must have adequate cardiac function(no cardiac disease, LVEF≥40% ), adequate pulmonary function as indicated by room air oxygen saturation of >94%, and adequate renal function(Cr≤133umol/L).
9. No other serious diseases(autoimmune disease, immunodeficiency etc.).
10. No other tumors.
11. Patients volunteer to participate in the research.
12. Patients with history of allogeneic stem cell transplantation are eligible if at least 100 days post-transplant, if there is no evidence of active GVHD and no longer taking immunosuppressive agents for at least 30 days prior to trial.

Exclusion Criteria:

1. KPS<50.
2. Patients are allergic to cytokines.
3. Central nervous system leukemia within 28 days.
4. Uncontrolled active infection.
5. Acute or chronic GVHD.
6. Treated with T cell inhibitor.
7. Pregnancy and nursing females.
8. HIV/HBV/HCV Infection.
9. Other situations we think improper for the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Antitumor Effects | Every 3 months post treatment up to 24 months
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

SECONDARY OUTCOMES:
Survival time of Anti-CD19 Anti-CD20 CAR T cells in vivo. | 3 years
  To evaluate the presence of circulating CAR T cells with flow cytometry and real time PCR in patient blood.
Adverse events of each patient. | 3 years
  Determine the toxicity profile of the CD19 CD20 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: li gangyi, Study Chair — Beijing Doing Biomedical Co., Ltd.
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China

IPD SHARING:
Plan to Share IPD: No